CLINICAL TRIAL: NCT04721925
Title: A Social Media Intervention for High-intensity Drinking in a National Sample of Emerging Adults
Brief Title: A Social Media Intervention for Risky Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Erin Bonar, Associate Professor of Psychiatry, Medical School and Adjunct Associate Professor of Psychology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00162416; R34AA027272-02 (NIH)
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Drinking Behavior
MeSH Terms: conditions — Drinking Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Link to an educational website about alcohol; link to resources.
- Social media messaging (Experimental): Health coaching via social media for 8 weeks
  Interventions: Behavioral: Social media messaging

INTERVENTIONS:
Behavioral: Social media messaging — A motivational interviewing-based intervention delivered via private health coaching on social media for 8 weeks.
  Arms: Social media messaging

SUMMARY:
This study is being completed to pilot prevention methods to promote wellness and reduce risky behaviors, including the use of substances such as alcohol and other drugs. This study will help the study team learn about ways of delivering this information that is both appealing and helpful to young adults.

ELIGIBILITY:
Inclusion Criteria:

* Reside in the United States of America (USA)
* Be able to read English, view, and click on a social media advertisement.
* Self-reported past-month high-intensity drinking (HID)
* Regular Snapchat use (at least 3 days/week).

Exclusion Criteria:

* If they fail identity verification based on: 1) internet protocol address (IP), 2) survey time completion, 3) repeat attempts, and 4) survey responses.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bonar, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A baseline assessment occurred prior to randomization. If consented individuals did not complete the assessment they were not randomized and thus not included in the study.
Period: 2-Month Assessment
Arm/Group | Control Group | Social Media Messaging
Started | 52 | 50
Completed (Completed 2 Month Assessment) | 47 | 47
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 3
Period: 4-Month Assessment
Arm/Group | Control Group | Social Media Messaging
Started | 52 | 50
Completed (Completed 4-Month Assessment) | 49 | 44
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Social Media Messaging | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (2.0) | 21.0 (2.0) | 20.9 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 27 | 25 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 27
  Not Hispanic or Latino | 35 | 40 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 34 | 32 | 66
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intervention Acceptability
Description: Study-specific acceptability rating completed by participants (% with a positive rating, higher % is better):
  Item wording: Overall, how did you feel about Snapchatting with the team? Response options: Disliked it a lot, Disliked it, Neutral, Liked it/Liked it a lot
  There are no statistical analyses because pre-registered primary outcomes are descriptive in nature.
Time Frame: 2 months
Population: 47 participants in the intervention group who completed a 2-month assessment. This measure is only reported among the intervention group arm because intervention acceptability can only be measured among those assigned to the intervention group. This measure would be irrelevant for the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Social Media Messaging
Number analyzed (Participants) | 47
Participants
  Disliked it a lot/Disliked it | 2
  Neutral | 5
  Liked it/Liked it a lot | 40

2. Primary Outcome: Feasibility of the Intervention (Engagement)
Description: % of participants engaging in the intervention (at least one reply) There are no statistical analyses because pre-registered primary outcomes are descriptive in nature.
Time Frame: During the 8 week intervention delivery period
Population: This measure is only reported among the intervention group arm because intervention acceptability can only be measured among those assigned to the intervention group. This measure would be irrelevant for the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Social Media Messaging
Number analyzed (Participants) | 50
Participants | 46

3. Primary Outcome: Feasibility of the Intervention (Completion)
Description: % of participants who remain connected to intervention account at 8 weeks (end of intervention) There are no statistical analyses because pre-registered primary outcomes are descriptive in nature.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Social Media Messaging
Number analyzed (Participants) | 50
Participants | 48

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up (approximately 4 months)
Arm/Group | Control Group | Social Media Messaging
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT04721925/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT04721925/ICF_000.pdf